CLINICAL TRIAL: NCT01508143
Title: A Comparative Study of Vaginal Misoprostol Two Dosing Regimen for First Trimester Pregnancy Termination in Patients Admitted at Bandarabbas in Shariati Hospital in 2009
Brief Title: Comparitive Study of Two Misoprostol Regimen in Early Pregnancy Termination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Mahboobi, Medical Doctor, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Misoprostol in termination
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Termination
Keywords: Abortion; Pregnancy; Termination; Misoprostol
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 400 microgram misoprostol (Experimental): 400 micrograms misoprostol each 6 hours for 8 dose
  Interventions: Drug: Misoprostol 400 micrograms
- 800 micrograms misoprostol (Active Comparator): 800 micrograms misoprostol each 12 hours for 4 dose
  Interventions: Drug: Misoprostol 800 micrograms

INTERVENTIONS:
Drug: Misoprostol 400 micrograms — Misoprostol 400 micrograms each 6 hours for 8 dose
  Other Names: Cytotec
  Arms: 400 microgram misoprostol
Drug: Misoprostol 800 micrograms — Misoprostol 800 micrograms each 12 hours for 4 doses
  Other Names: Cytotec
  Arms: 800 micrograms misoprostol

SUMMARY:
The aim of this study is to compare two misoprostol regimen in pregnancy termination.

DETAILED DESCRIPTION:
Studies on determining the optimal dosage for misoprostol in pregnancy termination are continuing and still there is no evidence for ideal misoprostol regimen for pregnancy termination. The aim of this study is to compare two misoprostol regimen in pregnancy termination.

ELIGIBILITY:
Inclusion Criteria:

* All women who were candidates for early pregnancy termination because of fetal death or other medical conditions
* Before 14th week of gestation calculated according LMP or first trimester sonography

Exclusion Criteria:

* Chorioamnionitis
* Hypersensitivity to prosstaglandins
* Past medical history of cardiovascular, kidney or liver or lung diseases
* Positive history for uterus pathologies
* suspicious to extra-uterus pregnancy
* sign and symptoms of uterus infection
* Molar pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Abortion | 48 hours after treatment
  After 48 hours after treatment each patient is assessed for abortion. Patients are devided into three groups including complete, partial or no abortion.

SECONDARY OUTCOMES:
Duration of abortion | Form the begining of treatment to complete abortion
  Duration of abortion Form the begining of treatment to complete abortion
Adverse Effects | 48 hours after treatment
  including nausea, vomiting, fever and chill, diarhea, abdominal cramp, skin rash
Need for surgery | 48 hours after treatment
  Dilatation & cartage

CONTACTS AND LOCATIONS:
Locations (1):
- Hormozgan University of Medical Sciences, Bandar Abbas, Hormozgan, Iran